CLINICAL TRIAL: NCT02173691
Title: A Multiple Dose Comparison of Tiotropium Inhalation Capsules, Salmeterol Inhalation Aerosol and Placebo in a Six-Month, Double-Blind, Double-Dummy, Safety and Efficacy Study in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety of Tiotropium Compared to Salmeterol and Placebo in Patients With Chronic Obstructive Bronchitis (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.137
Record Dates: First submitted 2014-06-20; First posted 2014-06-25 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Tiotropium (Experimental)
  Interventions: Drug: Tiotropium inhalation powder capsules; Drug: Placebo inhalation aerosol
- Salmeterol (Active Comparator)
  Interventions: Drug: Salmeterol inhalation aerosol; Drug: Placebo inhalation powder capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo inhalation aerosol; Drug: Placebo inhalation powder capsules

INTERVENTIONS:
Drug: Tiotropium inhalation powder capsules
  Arms: Tiotropium
Drug: Salmeterol inhalation aerosol
  Arms: Salmeterol
Drug: Placebo inhalation aerosol
  Arms: Placebo; Tiotropium
Drug: Placebo inhalation powder capsules
  Arms: Placebo; Salmeterol

SUMMARY:
The objective of this study is to compare the long-term (six month) bronchodilator efficacy and safety of tiotropium inhalation capsules, salmeterol inhalation aerosol and placebo inpatients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years.
* A diagnosis of relatively stable, moderate to severe COPD with:

  * Screening FEV1 ≤ 60% of predicted normal value (calculated according to European Community for Coal and Steel (ECCS) criteria and screening FEV1/FVC ≤ 70%
* Smoking history ≥ 10 pack-years (a pack-year is 20 cigarettes per day for one year or equivalent)
* Ability to be trained in the proper use of the HandiHaler® device and Metered Dose Inhaler (MDI).
* Ability to perform all study related tests including the Shuttle Walking Test, acceptable pulmonary function tests, including Peak expiratory flow rate (PEFR) measurements, and maintenance of diary card records.
* Ability to give written informed consent in accordance with Good Clinical Practice and local regulations.

Exclusion Criteria:

* Clinically significant diseases other than COPD.
* Patients with clinically relevant abnormal baseline haematology, blood chemistry or urinalysis, if the abnormality defines a disease listed as an exclusion criterion, will be excluded.
* All patients with a serum glutamic oxaloacetic transaminase (SGOT) > 80 IU/L, serum glutamic pyruvic transaminase (SGPT) > 80 IU/L, bilirubin >2.0 mg/dL or creatinine > 2.0 mg/dL will be excluded regardless of clinical condition.
* A recent history (i.e., one year or less) of myocardial infarction.
* Any cardiac arrhythmia requiring drug therapy or hospitalisation for heart failure within the past three years.
* Inability to abstain from regular daytime use of oxygen therapy for more than 1 hour per day.
* Known active tuberculosis.
* History of cancer within the last five years (excluding basal cell carcinoma)
* History of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis.
* Patients who have undergone thoracotomy with pulmonary resection.
* Any upper respiratory infection in the past six weeks prior to the screening visit or during the run-in period.
* Current participation in a pulmonary rehabilitation programme or completion of a pulmonary rehabilitation programme in the six week prior to the screening visit.
* Known hypersensitivity to anticholinergic drugs, salmeterol, or any of the components of the lactose powder capsule or MDI delivery systems.
* Known symptomatic prostatic hypertrophy or bladder neck obstruction.
* Patients with known narrow-angle glaucoma.
* Current treatment with cromolyn sodium or nedocromil sodium.
* Current treatment with antihistamines (H1 receptor antagonists).
* Oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisolone per day or 20 mg every other day.
* Current use of β-blocker medication.
* Current treatment with monoamine oxidase inhibitors or tricyclic antidepressants.
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception.
* Patients with a history of asthma, allergic rhinitis or atopy or who have a total blood eosinophil count > 600mm3.
* History of and/or active significant alcohol or drug abuse.
* Concomitant or recent use of an investigational drug within one month or six half lives (whichever is greater) prior to the screening visit.
* Changes in the pulmonary therapeutic plan within the six weeks prior to the screening visit.
* Inability to comply with the medication restrictions specified in Section 4.2 of the trial protocol

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 1999-02; Primary Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Trough forced expiratory volume in one second (FEV1) response | 6 months
Transition Dyspnoea Index (TDI) focal score | 6 months

SECONDARY OUTCOMES:
Average FEV1 response | 30 and 60 min prior to and 30 and 60 min, 2 and 3 h post treatment on day 1, week 2, 8, 16, 24
Peak FEV1 response | 30 and 60 min prior to and 30 and 60 min, 2 and 3 h post treatment on day 1, week 2, 8, 16, 24
Trough FVC (forced vital capacity) response | 30 and 60 min prior to and 30 and 60 min, 2 and 3 h post treatment on day 1, week 2, 8, 16, 24
Average FVC (forced vital capacity) response | 30 and 60 min prior to and 30 and 60 min, 2 and 3 h post treatment on day 1, week 2, 8, 16, 24
Peak FVC (forced vital capacity) response | 30 and 60 min prior to and 30 and 60 min, 2 and 3 h post treatment on day 1, week 2, 8, 16, 24
Individual FEV1 measurement | Day 1, weeks 2, 8, 16, 24
Individual FVC measurement | Day 1, weeks 2, 8, 16, 24
Patient peak expiratory flow rates (PEFR) twice daily | 27 weeks
Physician's global evaluation on an 8-point-scale | 27 weeks
COPD symptom scores (wheezing, shortness of breath, coughing and tightness of chest) | 27 weeks
Amount of salbutamol therapy used during the treatment period | 27 weeks
Number and length of exacerbations of COPD | 27 weeks
Number and length of hospitalizations for respiratory disease | 27 weeks
Changes from baseline in St. George's Hospital Respiratory Questionnaire (SGRQ) | Day 1, week 8, 16, 24 and 27
Changes from baseline in Mahler Dyspnoea Index (Baseline Dyspnoea Index /Transitional Dyspnoea Index (BDI/TDI)) | Baseline, week 8, 16, 24, 27
Health resource utilisation | 27 weeks
Patient preference measures | Day 1 and week 24
  patient satisfaction questionnaire score
Changes from baseline in Shuttle walking tests (SWT) and Borg dyspnea score | Day 1, week 8, 16, 24, 27
Occurrence of Adverse Events | 27 weeks
Changes from baseline in pulse rate and blood pressure in conjunction with spirometry | baseline, Day 1, week 2, 8, 16 and 24
Changes from baseline in physical examination and ECG | baseline and week 24
Changes from baseline in laboratory tests | baseline and week 24